CLINICAL TRIAL: NCT00057499
Title: Autoantigen Vaccination in Human Type 1 Newly Diagnosed Diabetes Mellitus
Brief Title: Evaluation of a Diabetes Vaccine in Newly Diagnosed Diabetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAIT ITN012AI; DAIT BD012
Record Dates: First submitted 2003-04-03; First posted 2003-04-04 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Insulin-dependent Diabetes Mellitus; Diabetes Mellitus
Keywords: Juvenile diabetes; Diabetes; Insulin; Vaccine; Type 1 Diabetes; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IBC-VS01 vaccine (Experimental): IBC-VS01 vaccine is administered twice.
  Interventions: Biological: IBC-VS01
- Control Group (Placebo Comparator): IBC-VS01 placebo is administered twice
  Interventions: Biological: IBC-VS01 placebo

INTERVENTIONS:
Biological: IBC-VS01 — IBC-VS01
  Arms: IBC-VS01 vaccine
Biological: IBC-VS01 placebo — IBC-VS01 placebo
  Arms: Control Group

SUMMARY:
Insulin dependent diabetes mellitus (also called type 1 diabetes mellitus or T1DM) is caused by the destruction of insulin-producing cells in the pancreas. People with T1DM do not produce enough insulin, which is necessary for proper regulation of blood sugar levels.

T1DM is an autoimmune disease. An autoimmune disease is a disease in which the body's immune system attacks the body itself. In addition to regulating blood sugar, insulin may have the ability to protect cells in the pancreas from attack by the immune system. This study will evaluate whether an insulin-based vaccine can protect cells from autoimmune destruction.

Study hypothesis: IFA-enhanced human insulin B-chain vaccination will lead to the arrest or slowing of the ongoing autoimmunity, and this will result in an appreciable difference in functioning B cell mass compared to the placebo treated group by the end of the study.

DETAILED DESCRIPTION:
The vaccine in this study, IBC-VSO1, is a synthetic, metabolically inactive form of insulin designed to prevent pancreatic beta-cell destruction. It does not cause fluctuations in blood sugar. This study will evaluate whether the vaccine protects against autoimmune attack at the onset of T1DM, before pancreas function has deteriorated. This experimental treatment must occur early because 60% to 85% of beta-cells are already destroyed by the time of T1DM diagnosis. If beta-cell destruction can be halted, a prolonged remission period after diagnosis may occur, with a subsequent delay in diabetes-related complications.

Participants must have been diagnosed with T1DM for no more than 3 months at the time of enrollment in this study. Participants will be randomly assigned to either a vaccine group or a control group. Participants in the vaccine group will receive one injection of IBC-VS01; participants in the control group will receive a placebo. Participants will then be monitored for 2 years. Participants will have ten follow-up visits, which will include blood tests for immunological and genetic analysis. Throughout the study, metabolic tests will also be performed to measure the remaining capacity of self insulin production of the body.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 1 diabetes mellitus within 3 months prior to study entry
* Positive for IAA, GAD65, or IA2 antibodies OR positive for GAD65 or IA2 antibodies after 2 weeks of starting insulin treatment

Exclusion Criteria:

* History of treatment with any oral hypoglycemic agent for more than 3 months
* Ongoing use of medications known to influence glucose tolerance
* History of immunosuppressive or steroid therapy for more than 3 months within the 2 years prior to study entry
* Severe active liver, heart, kidney, or immunodeficiency disease that may limit life expectancy or may require immunosuppression during the study
* Prior complications related to routine vaccinations
* Prior participation in a trial for prevention of type 1 diabetes mellitus. Individuals who are known to have been in the placebo arm of a completed prevention trial are not excluded.
* Any condition that may interfere with a participant's ability to comply with the study
* Pregnancy or planned pregnancy within the time frame of the study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2003-03; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Clinical endpoints including adverse events, local reactions, routine physical exams, insulin dose, and laboratory tests | Throughout study

SECONDARY OUTCOMES:
C-peptide levels in response to mixed meal tolerance test | Throughout study
HbA1c, GAD65Ab, IAA, IA2Ab, GAD65Ab isotypes | Throughout study
CD4- and CD8- Va24JaQ+ | Throughout study
T cells' secretion of IL-4 and Interferon (IFN)-gamma | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Tihamer Orban, MD, Principal Investigator — Joslin Diabetes Center
Locations (2):
- United States (2):
  - Children's Hospital, Boston, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Data access is provided to the public in : 1.) the Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts that also provides data analysis tools available to researchers; and 2.) TrialShare, the Immune Tolerance Network (ITN) portal.

REFERENCES:
- [Result] Orban T, Farkas K, Jalahej H, Kis J, Treszl A, Falk B, Reijonen H, Wolfsdorf J, Ricker A, Matthews JB, Tchao N, Sayre P, Bianchine P. Autoantigen-specific regulatory T cells induced in patients with type 1 diabetes mellitus by insulin B-chain immunotherapy. J Autoimmun. 2010 Jun;34(4):408-15. doi: 10.1016/j.jaut.2009.10.005. PMID 19931408
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) website — https://www.niaid.nih.gov/about/dait
- See also: Immune Tolerance Network (ITN) website — http://www.immunetolerance.org
- Available data/document: Individual Participant Data Set: SDY568 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY568 — ImmPort study identifier is SDY568.
- Available data/document: Study summary, -schematic, -design, medications,-demographics, - lab tests, -study files: SDY568 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY568 — ImmPort study identifier is SDY568.
- Available data/document: Individual Participant Data Set: ITN012AI — http://www.itntrialshare.org/project/Studies/ITN012AIPUBLIC/Study%20Data/begin.view? — TrialShare is the Immune Tolerance Network (ITN) portal that makes data from the consortium's clinical trials publicly available without charge. Creating an account for ITN TrialShare is free and allows for searching studies of interest.
- Available data/document: Study protocol synopsis, -navigator, -schedule of events,-data &reports, -specimens et al.: ITN012AI — http://www.itntrialshare.org/project/Studies/ITN012AIPUBLIC/Study%20Data/begin.view? — TrialShare is the Immune Tolerance Network (ITN) portal that makes data from the consortium's clinical trials publicly available without charge. Creating an account for ITN TrialShare is free and allows for searching studies of interest.